CLINICAL TRIAL: NCT00732836
Title: Phase I Trial of Hepatic Arterial Infusion of Abraxane With a Pharmacokinetic Study in Advanced Solid Cancer Patients With Predominant Hepatic Metastases
Brief Title: Hepatic Arterial Infusion (HAI) of Abraxane
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: M.D. Anderson Cancer Center (Other)
Collaborators: National Comprehensive Cancer Network (Network)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2007-0857; NCI-2012-02124 (Registry Identifier: NCI CTRP)
Record Dates: First submitted 2008-08-08; First posted 2008-08-12 (Estimated); Last update posted 2016-02-05 (Estimated); Status verified 2016-02

CONDITIONS: Liver Cancer; Advanced Cancers; Solid Tumors
Keywords: Liver Cancer; Solid Cancer; Abraxane; nab paclitaxel; HAI abraxane; HAI; hepatic arterial infusion; hepatic metastases
MeSH Terms: conditions — Liver Neoplasms | interventions — Taxes; 130-nm albumin-bound paclitaxel; Albumin-Bound Paclitaxel

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- HAI Abraxane MTD (Experimental): Dose escalation beginning Day 1, Cycle 2 dose level 180 mg/m^2 for maximum tolerated dose (MTD) of Hepatic Arterial Infusion of Abraxane (HAI Abraxane) following same dose intravenous Abraxane in Cycle 1 of 21 day cycle.
  Interventions: Drug: HAI Abraxane; Procedure: Hepatic Artery Catheter; Drug: IV Abraxane
- HAI Abraxane Expansion (Experimental): HAI Abraxane dose expansion at MTD or dose level 3 (260 mg/m^2) if MTD not defined.
  Interventions: Drug: HAI Abraxane; Procedure: Hepatic Artery Catheter

INTERVENTIONS:
Drug: HAI Abraxane — Escalating doses (beginning dose 180 mg/m^2) starting Day 1, Cycle 2 and later via hepatic arterial infusion (HAI) following IV Abraxane in Day 1, Cycle 1 for 21 day cycles.
  Other Names: Nab Abraxane; Paclitaxel (protein-bound); Nab-paclitaxel; Abraxane; Coroxane; Capxol
Procedure: Hepatic Artery Catheter — On each day of treatment for Cycles 2-4, hepatic artery catheter placement completed by interventional radiology.
  Other Names: HAI
Drug: IV Abraxane — Intravenous (IV) Abraxane only in Cycle 1 (up to Dose Level 4 of 260 mg/m^2), infused over 60 minutes or 4 hours Day 1 of 21 day cycle.
  Other Names: Nab Abraxane; Paclitaxel (protein-bound); Nab-paclitaxel; Abraxane; Coroxane; Capxol
  Arms: HAI Abraxane MTD

SUMMARY:
The goal of this clinical research study is find the highest tolerated dose of Abraxane (nab-paclitaxel) that can be given directly into the liver of patients with advanced cancer that has spread to the liver.

DETAILED DESCRIPTION:
The Study Drug:

Nab-paclitaxel is designed to block cancer cells from dividing, which may cause the cells to die.

Giving nab-paclitaxel directly into the liver may allow a higher dose of the drug to be given, while avoiding some of the side effects that occur when high doses of chemotherapy are given other ways (for example, by vein into an arm).

Study Drug Dose Level:

If you are found to be eligible to take part in this study, you will be assigned to a study group based on when you joined this study. Up to 9 groups of 6 participants will be enrolled in Part 1 of the study, and up to 18 participants will be enrolled in Part 2. If you are enrolled in Part 1, the dose of the study drug you receive will depend on when you joined this study. The first group of participants will receive the lowest dose level of the study drug. Each new group will receive a higher dose of the study drug than the group before it, if no intolerable side effects were seen. This will continue until the highest tolerable dose of the study drug is found. If you are enrolled in Part 2, you will receive the study drug at the highest dose that was tolerated in the Part 1 portion.

Study Drug Administration:

The study drug will be given on Day 1 of "cycles" that are 21 days long. In Cycle 1 only, some participants may receive the study drug through a vein in their arm. The infusion will last 60 minutes. In Cycles 2 and later, you will receive the study drug through a catheter (a thin plastic tube). Each time the catheter is placed, you will be admitted to the hospital.

The doctor who performs the catheter placement procedure will explain it to you in more detail, and you will be asked to sign a separate consent form that describes the procedure and its risks in more detail.

You will be taken to the Interventional Radiology area, and the catheter will be placed in a blood vessel in your groin area, on the right side of your body. The catheter will be advanced to the liver. The catheter will be carefully taped in order to prevent it from moving or coming out while you are receiving the study drug. You will be on bedrest for the entire time that the catheter is in place.

After having the catheter inserted, you will be taken to the Nuclear Medicine area, and a test called "flow study" will be performed in order to confirm that the catheter is in the right place. The doctor who performs this test will explain it to you in more detail, and you will be asked to sign a separate consent form that describes the procedure and its risks in more detail.

After you return to your room, you will receive the study drug through the catheter over 60 minutes or 4 hours, depending on when you enroll. You will be asked to lie flat on your back while receiving the study drug.

The catheter will be removed by someone experienced in the procedure. It will be removed right after your study drug dose is complete. While the catheter is being removed, the study staff will apply pressure to your groin area for 15 minutes in order to stop the bleeding.

You will repeat this procedure once every 21 days. The catheter will be placed and removed each time.

Study Procedures and Tests:

Once a week, including before each dose of the study drug, blood (about 2 teaspoons) will be drawn for routine tests. These blood draws can be done at M. D. Anderson or somewhere else, if there is a place that is more convenient for you.

Once during each cycle (on a day when you are already in clinic), you will have a physical exam, including measurement of height, weight, and vital signs. Urine will be collected for routine tests.

At the end of every 3 cycles, you will have scans performed (the same type of scans as at screening) to check the status of the disease. If the study doctor feels it is appropriate, you may have blood drawn (about 1 teaspoon) to look for tumor markers.

Blood Testing for Research Purposes:

In Cycles 1 and 2, additional blood will be drawn for pharmacokinetic (PK) testing. PK testing measures the amount of study drug in the body at different time points. For participants receiving the study drug over 60 minutes, this blood (about 1 teaspoon each time) will be drawn on Day 1 (before you receive the study drug and at 5, 10, 20 and 40 minutes after the start of the dose, and then at 1, 1½, 2, 3, 4, and 6 hours after the start of the dose). Blood will also be drawn on Day 2 (24 hours after the start of the dose).

For participants receiving the study drug over 4 hours, this blood (about 1 teaspoon each time) will be drawn on Day 1 (before you receive the study drug and at 30 minutes after the start of the dose, and then at 1, 2, 3, 4, 4 ½, 5, 6, 7, and 9 hours after the start of the dose). Blood will also be drawn on Day 2 (24 hours after the start of the dose).

Length of Study Participation:

You will continue to receive the study drug once every 21 days. If the disease gets worse or intolerable side effects occur, you will be taken off the study drug.

End-of-Study Visit:

After your last dose of the study drug, you will have an end-of-study visit. At this visit, the following procedures will be performed:

* You will have a physical exam, including measurement of weight and vital signs.
* Blood (about 2 tablespoons) and urine will be collected for routine tests.
* To check the status of the disease, you will have scans performed (the same types of scans that you had before).
* If the study doctor feels it is appropriate, you may have blood drawn (about 1 teaspoon) to look for tumor markers.

This is an investigational study. Nab-paclitaxel is commercially available and FDA approved for use in breast cancer and for "systemic" use only. Systemic therapies affect the body as a whole. It is investigational to give nab-paclitaxel directly into the liver and to give it to patients with advanced cancer. At this time, giving it directly into the liver of patients with advanced cancer is only being done in research.

Up to 56 patients will take part in this study. All will be enrolled at M. D. Anderson.

ELIGIBILITY:
Inclusion Criteria:

1. Pathologically confirmed diagnosis of advanced malignancy and liver involvement as predominant site of metastasis.
2. An Eastern Cooperative Oncology Group (ECOG) performance status of 0-2
3. Adequate end-organ function as follows: Absolute neutrophil count (ANC) > or = 1500/mm3, Platelets > or = 100,000/mm3, Creatinine < or = 2.0 mg/dL or the calculated Glomerular filtration rate (GFR) > or = 40 mL/min if Creatinine > 2.0 mg/dL, ALT < or = 5 times upper limits of normal, Hb > 9.0 and Bilirubin < or = 2.0 mg/dL.
4. Refractory to standard cancer therapy or who have no conventional therapy that produces a complete response rate of at least 10% or an increase in survival of at least 3 months.
5. Ability to fully comprehend and willingness to sign the Institutional Review Board (IRB) approved informed consent
6. Full recovery from any previous therapy and ability to receive cytotoxic agents.
7. Patient is 18 years of age or older

Exclusion Criteria:

1. Clinically significant ascites.
2. Pregnant or breastfeeding females. Women of childbearing potential should be advised to avoid becoming pregnant and men to not father a child while receiving treatment. Women of childbearing potential must have a negative pregnancy test.
3. Hypersensitivity to Abraxane
4. Untreatable bleeding diathesis
5. Evidence of portal vein thrombosis and clinically significant peripheral vascular disease
6. Neuropathy of grade 2 or higher
7. A known history of central nervous system (CNS) metastasis unless the patients are neurologically stable after treatment with surgery and/or radiation therapy
8. If the patient progressed on abraxane previously they will not be eligible for the dose escalation portion or the PK studies only. These patients can be included in the dose expansion portion of the trial.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 64 (Actual)
Dates: Start 2008-06; Primary Completion 2016-01 (Actual); Study Completion 2016-01 (Actual)

PRIMARY OUTCOMES:
Maximum Tolerated Dose (MTD) of HAI Abraxane | Assessments every 3 week cycle (21 days)
  MTD is highest dose level in which 6 patients with at most 1 patient experiencing a dose limiting toxicity (DLT). Dose escalation continues until DLT is defined or until dose level 4 is completed. DLT defined during first cycle of treatment.

CONTACTS AND LOCATIONS:
Overall Officials: Siqing Fu, MD, PHD, Principal Investigator — M.D. Anderson Cancer Center
Locations (1):
- University of Texas MD Anderson Cancer Center, Houston, Texas, United States

REFERENCES:
- [Derived] Siqing F, Culotta KS, Falchook GS, Hong DS, Myers AL, Zhang YP, Naing A, Janku F, Hou MM, Kurzrock R. Pharmacokinetic evaluation of nanoparticle albumin-bound paclitaxel delivered via hepatic arterial infusion in patients with predominantly hepatic metastases. Cancer Chemother Pharmacol. 2016 Feb;77(2):357-64. doi: 10.1007/s00280-015-2946-x. Epub 2015 Dec 23. PMID 26698868
- See also: University of Texas MD Anderson Cancer Center Website — http://www.mdanderson.org